CLINICAL TRIAL: NCT02317861
Title: A Phase 2a, Randomized, Open-Label, Single-Site Study to Evaluate the Pharmacodynamic Effects and Safety of RDEA3170 Administered in Combination With Febuxostat Compared to RDEA3170 Administered Alone and Febuxostat Administered Alone, Respectively in Japanese Adult Male Subjects With Gout or Asymptomatic Hyperuricemia
Brief Title: A PD/Safety Study of RDEA3170 in Combination With Febuxostat for Treating Gout or Asymptomatic Hyperuricemia Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D5491L00001; RDEA3170-205 (Other: Ardea Biosciences, Inc.)
Record Dates: First submitted 2014-12-09; First posted 2014-12-17 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Gout and Asymptomatic Hyperuricemia
MeSH Terms: conditions — Gout | interventions — verinurad; Febuxostat; Benzbromarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): The half of patients randomized to this cohort will be dosed in the order of Febuxostat 10mg, RDEA3170 2.5 mg + Febuxostat 10mg, RDEA3170 2.5 mg + Febuxostat 20mg, and Febuxostat 20mg. The other half will be dosed in the reverse order.
  Interventions: Drug: RDEA3170; Drug: Febuxostat
- Cohort 2 (Experimental): The half of patients randomized to this cohort will be dosed in the order of Febuxostat 10mg, RDEA3170 5 mg + Febuxostat 10mg, RDEA3170 5 mg + Febuxostat 20mg, and Febuxostat 20mg. The other half will be dosed in the reverse order.
  Interventions: Drug: RDEA3170; Drug: Febuxostat
- Cohort 3 (Experimental): The half of patients randomized to this cohort will be dosed in the order of Febuxostat 20mg, RDEA3170 5 mg + Febuxostat 20mg, RDEA3170 5 mg + Febuxostat 40mg, and Febuxostat 40mg. The other half will be dosed in the reverse order.
  Interventions: Drug: RDEA3170; Drug: Febuxostat
- Cohort 4 (Experimental): The half of patients randomized to this cohort will be dosed in the order of Febuxostat 20mg, RDEA3170 10 mg + Febuxostat 20mg, RDEA3170 10 mg + Febuxostat 40mg, and Febuxostat 40mg. The other half will be dosed in the reverse order.
  Interventions: Drug: RDEA3170; Drug: Febuxostat
- Cohort 5 (Experimental): RDEA3170 2.5mg, RDEA3170 5mg, RDEA3170 10mg, RDEA3170 15mg
  Interventions: Drug: RDEA3170
- Cohort 6 (Experimental): The half of patients randomized to this cohort will be dosed in the order of Benzbromarone 50 mg, Febuxostat 10mg+RDEA3170 2.5 mg, then Febuxostat 20mg+RDEA3170 5 mg. The other half will be dosed in the order of Febuxostat 10mg+RDEA3170 2.5 mg, Febuxostat 20mg+RDEA3170 5 mg, then Benzbromarone 50mg.
  Interventions: Drug: RDEA3170; Drug: Febuxostat; Drug: Benzbromarone

INTERVENTIONS:
Drug: RDEA3170 — Oral Treatment
Drug: Febuxostat — Oral Treatment
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 6
Drug: Benzbromarone — Oral Treatment
  Arms: Cohort 6

SUMMARY:
The purpose of this study is to explore the pharmacodynamics (PD), pharmacokinetics (PK), safety, and tolerability of multiple doses of RDEA3170 administered in combination with febuxostat compared to RDEA3170 administered alone and febuxostat administered alone in Japanese adult male subjects with gout or asymptomatic hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* Screening serum uric acid level ≥ 8 mg/dL;
* Body weight ≥ 50 kg and a body mass index (BMI) ≥ 18 and ≤ 40 kg/m2;
* Free of any clinically significant disease or medical condition, per the Investigator's judgment.

Exclusion Criteria:

* History or suspicion of kidney stones;
* Diagnosis of benign prostatic hypertrophy (BPH) or neurogenic bladder or evidence of BPH/neurogenic bladder such as thin urinary stream or difficulty in urination;
* An estimated creatinine clearance < 60 mL/min calculated by the Cockcroft-Gault formula;
* QTcF interval (QT interval corrected for heart rate using Fridericia's formula) > 450 msec at Screening;
* Receiving strong or moderate Cytochrome P450 (CYP) 3A inhibitors or p-glycoprotein inhibitors, or digoxin

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Serum uric acid level | baseline and day 7 on each treatment
  % change per treatment will be compared.
Change in Urinary excretion of uric acid | baseline and day 7 on each treatment
  Timed urinary uric acid excretion per treatment will be compared
Renal clearance of uric acid | baseline and day 7 on each treatment
  Renal clearance of uric acid will be calculated.
Fractional excretion of uric acid | baseline and day 7 on each treatment
  Fractional excretion and renal clearance of uric acid will be calculated.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 , 24 hours post-dose on each treatment
  To assess multiple-dose PK of RDEA3170 and febuxostat alone or in combination treatment.
Time to reach maximum concentration (tmax) | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 , 24 hours post-dose on each treatment
  To assess multiple-dose PK of RDEA3170 and febuxostat alone or in combination treatment.
Area under the concentration-time curve (AUC) | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 , 24 hours post-dose on each treatment
  To assess multiple-dose PK of RDEA3170 and febuxostat alone or in combination treatment.
Half life (t1/2) | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 , 24 hours post-dose on each treatment
  To assess multiple-dose PK of RDEA3170 and febuxostat alone or in combination treatment.
Incidence of adverse events | Day 1 and Day 7 on each treatment
  To evaluate the safety and tolerability of febuxostat alone, RDEA3170 alone and RDEA3170 administered in combination of febuxostat and febuxostat in combination of RDEA3170
Changes in hematology, serum chemistry, coagulation, electrocardiogram and urinalysis parameters | Day 1 and Day 8 on each treatment
  To evaluate the safety and tolerability of febuxostat alone, RDEA3170 alone and RDEA3170 administered in combination of febuxostat and febuxostat in combination of RDEA3170
Changes in vital signs and physical examination findings | Day 1 and Day 8 on each treatment
  To evaluate the safety and tolerability of febuxostat alone, RDEA3170 alone and RDEA3170 administered in combination of febuxostat and febuxostat in combination of RDEA3170
Incidence of adverse events | Day 42 of the study as follow up
  To evaluate the safety and tolerability of febuxostat alone, RDEA3170 alone and RDEA3170 administered in combination of febuxostat and febuxostat in combination of RDEA3170
Changes in hematology, serum chemistry, coagulation, electrocardiogram and urinalysis parameters | Day 42 of the study as follow up
  To evaluate the safety and tolerability of febuxostat alone, RDEA3170 alone and RDEA3170 administered in combination of febuxostat and febuxostat in combination of RDEA3170
Changes in vital signs and physical examination findings | Day 42 of the study as follow up
  To evaluate the safety and tolerability of febuxostat alone, RDEA3170 alone and RDEA3170 administered in combination of febuxostat and febuxostat in combination of RDEA3170

OTHER OUTCOMES:
Change in Urinary pH | baseline and day 7 on each treatment
  To evaluate the relationship between the doses of uralyt and urinary pH under the administration of RDEA3170.
Deoxyribonucleic acid polymorphism | Day 1 of the study as randomization
  To collect and store deoxyribonucleic acid (DNA) for future exploratory research.
Change in Serum uric acid level | Baseline and day 7 on each treatment for cohort 6
  % change per treatment will be compared.
Change in Urinary excretion of uric acid | Baseline and day 7 on each treatment for cohort 6
  Timed urinary uric acid excretion per treatment will be compared.
Renal clearance of uric acid | Baseline and day 7 on each treatment for cohort 6
  Renal clearance of uric acid will be calculated.
Fractional excretion of uric acid | Baseline and day 7 on each treatment for cohort 6
  Fractional excretion and renal clearance of uric acid will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Fukuoka, Japan

REFERENCES:
- [Derived] Rekic D, Johansson S, Leander J. Higher Febuxostat Exposure Observed in Asian Compared with Caucasian Subjects Independent of Bodyweight. Clin Pharmacokinet. 2021 Mar;60(3):319-328. doi: 10.1007/s40262-020-00943-6. Epub 2020 Sep 19. PMID 32951150
- [Derived] Shiramoto M, Liu S, Shen Z, Yan X, Yamamoto A, Gillen M, Ito Y, Hall J. Verinurad combined with febuxostat in Japanese adults with gout or asymptomatic hyperuricaemia: a phase 2a, open-label study. Rheumatology (Oxford). 2018 Sep 1;57(9):1602-1610. doi: 10.1093/rheumatology/key100. PMID 29868853